CLINICAL TRIAL: NCT02566031
Title: A Randomized, Multicenter, Open-label, Parallel-group, 12-week Study to Assess the Efficacy and Safety of Switching From Tiotropium to QVA149 (Indacaterol Maleate/Glycopyrronium Bromide) in Symptomatic Mild to Moderate COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQVA149AKR01
Record Dates: First submitted 2015-08-10; First posted 2015-10-01 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: COPD
Keywords: COPD; open-label; QVA149; symptomatic; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate; indacaterol-glycopyrronium combination; Tiotropium Bromide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indacaterol and glycopyrronium (QVA149) (Experimental): QVA149 110/50 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDPPI) for 12 weeks
  Interventions: Drug: Indacaterol and glycopyrronium (QVA149)
- Tiotropium (Active Comparator): Tiotropium 18 μg capsules for inhalation delivered once daily via HandiHaler® device for 12 weeks
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Indacaterol and glycopyrronium (QVA149) — Capsules for inhalation delivered via SDDPI
  Arms: Indacaterol and glycopyrronium (QVA149)
Drug: Tiotropium — Capsules for inhalation delivered via HandiHaler® device
  Arms: Tiotropium

SUMMARY:
To demonstrate superiority of QVA149 (110/50 μg) once daily compared to tiotropium 18 μg once daily in terms of trough forced expiratory volume in 1 second (FEV1) (mean of 45 min and 15 min pre-dose) following 12 weeks of treatment in mild to moderate symptomatic COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COPD and post-bronchodilator FEV1 ≥ 50% of the predicted normal value and post-bronchodilator FEV1/FVC < 0.7 (COPD Grade 1 or 2 by severity of airflow limitation (GOLD 2015)
* Patients with CAT score ≥ 10 at Visit 0 and Visit 1.
* Patients who are on and have been on tiotropium monotherapy for the past 3 months.
* 0 or 1 COPD exacerbation in the previous 12 months (not leading to hospital admission).

Exclusion Criteria:

* Treatment with any inhaled corticosteroid (ICS) in the 3 months prior to Visit 1.
* COPD exacerbation between Visit 0 and 1.
* Patients with concomitant pulmonary disease
* Patients with a history of respiratory infection within 4 weeks prior to Visit 0.
* Prior or current diagnosis of asthma.
* Presence of any contraindication, warning, precaution, hypersensitivity to LABA and LAMA

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Novartis Investigative Site, Chuncheon, Gangwon-do
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Guri-si, Gyeonggi-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Jeju City
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Ulsan

REFERENCES:
- [Derived] Rhee CK, Park HY, Park JW, Lee JH, Kim TH, Lee SW, Jung JY, Kim S, Hwang YI, Jung KS. Efficacy and safety of indacaterol/glycopyrronium fixed-dose combination in mild-to-moderate COPD patients symptomatic on tiotropium in Korea: study protocol for a randomized controlled trial. Trials. 2017 Feb 22;18(1):80. doi: 10.1186/s13063-017-1800-3. PMID 28228162

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Started | 189 | 190
Completed | 169 | 178
Not Completed | 20 | 12
Not completed — Patient/guardian decision | 14 | 7
Not completed — Protocol deviation | 2 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium | Total
Number analyzed (Participants) | 189 | 190 | 379
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (8.08) | 69.0 (7.54) | 69.1 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 186 | 183 | 369
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 189 | 190 | 379
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume In One Second (FEV1) After 12 Weeks of Treatment
Description: Spirometry was performed according to internationally accepted standards. Trough FEV1 is defined as the mean of 45 minute and 15 minute pre-dose values.
Time Frame: Week 12
Population: The full analysis set (FAS) consisted of all randomized patients who received at least one dose of study treatment and have at least one evaluable post-baseline assessment.
  Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 177 | 184
Liters | 0.0668 (0.18097) | 0.0090 (0.18487)
Statistical Analysis 1: Comparison: Indacaterol and Glycopyrronium (QVA149) vs Tiotropium; Test type: Superiority; p = 0.0129, ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [0.011 to 0.093]

2. Secondary Outcome: Trough Forced Expiratory Volume In One Second (FEV1) After 4 Weeks of Treatment
Description: Spirometry was performed according to internationally accepted standards. Trough FEV1 was defined as the mean of 45 minute and 15 minute pre-dose values.
Time Frame: mean of 45 min and 15 min pre-dose week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 177 | 184
Liters
  -45min: number analyzed (Participants) | 175 | 179
  -45min | 0.087 (0.2386) | 0.026 (0.1626)
  -15min: number analyzed (Participants) | 174 | 179
  -15min | 0.077 (0.2298) | 0.024 (0.1567)
Statistical Analysis 1: Comparison: Indacaterol and Glycopyrronium (QVA149) vs Tiotropium; -45 min; Test type: Superiority; p = 0.0058, ANCOVA; Mean Difference (Net) = 0.06, 95% CI 2-sided [0.017 to 0.098]
Statistical Analysis 2: Comparison: Indacaterol and Glycopyrronium (QVA149) vs Tiotropium; -15min; Test type: Superiority; p = 0.0161, ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [0.009 to 0.091]

3. Secondary Outcome: Baseline Transitional Dyspnea Index (TDI) Focal Score
Description: A trained assessor interviewed the patient and graded the degree of impairment due to dyspnea (difficulty breathing). TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort and captures changes from baseline. TDI captures changes from baseline, each domain is scored from -3=major deterioration to 3=major improvement to give an overall TDI focal score of -9 to 9. Higher numbers indicate a better score.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 177 | 184
Score | 0.77 (1.735) | 0.61 (1.534)
Statistical Analysis 1: Comparison: Indacaterol and Glycopyrronium (QVA149) vs Tiotropium; Test type: Superiority; p = 0.0767, ANCOVA; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.033 to 0.646]

4. Secondary Outcome: Number of Participants With Change From Baseline on Total Score of COPD Assessment Test (CAT)
Description: Total score of COPD Assessment Test (CAT) will be measured at week 12. This questionnaire is completed by the patient. The score ranges from 0-40 where higher scores represent worse health status. Mild: Score = 0 - 10, Moderate: Score = 11 - 20, Severe: Score = 21 - 30, Very Severe: Score = 31 - 40. The CAT total score was the sum of 8 item scores (each ranging from 0 to 5). If 1 or 2 items were missing, they were replaced with the mean of the completed items. If 3 or more items were missing, the CAT total score was set missing
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 177 | 184
Number of participants
  Mild | 62 | 54
  Moderate | 92 | 101
  Severe | 15 | 22
  Very severe | 0 | 1
  Missing | 8 | 6
Statistical Analysis 1: Comparison: Indacaterol and Glycopyrronium (QVA149) vs Tiotropium; Test type: Superiority; p = 0.1008, ANCOVA; Mean Difference (Net) = -0.81, 95% CI 2-sided [-1.77 to 0.16]

5. Secondary Outcome: Daily Rescue Medication Use (Number of Puffs)
Description: The total number of puffs of rescue medication used over the last 24 hours will be recorded in the patient diary in the morning. The total number of puffs of rescue medication per day over the full 12 weeks will be calculated and divided by the total number of days with non-missing rescue medication data to derive the mean daily number of puffs of rescue medication taken for the patient. The mean daily number of puffs of rescue medication used over 12 weeks will be summarized by treatments
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Indacaterol and Glycopyrronium (QVA149) | Tiotropium
Number analyzed (Participants) | 177 | 184
Puffs/day | 1.7 (0.92) | 1.8 (1.28)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Groups:
- Indacaterol and Glycopyrronium (QVA149: QVA149 110/50 μg capsules for inhalation delivered once daily via single-dose dry powder inhaler (SDPPI) for 12 weeks
- Total: Total
Arm/Group | Indacaterol and Glycopyrronium (QVA149 | Tiotropium | Total
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/188 | 0/377
Serious Adverse Events (participants affected / at risk) | 8/189 | 3/188 | 11/377
Other Adverse Events (participants affected / at risk) | 12/189 | 9/188 | 21/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium (QVA149 (N=189) | Tiotropium (N=188) | Total (N=377)
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol and Glycopyrronium (QVA149 (N=189) | Tiotropium (N=188) | Total (N=377)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT02566031/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02566031/SAP_001.pdf